CLINICAL TRIAL: NCT01999413
Title: Pilot Study of the Efficacy and Tolerance of the Adjunction of a Fish Oil Emulsion to Daunorubicin and Cytarabine Chemotherapy for the Treatment of Acute MYeloblastic Leukemia of Younger Patients With High-risk Cytogenetics
Brief Title: Pilot Study Efficacy and Tolerance Fish Oil Emulsion Daunorubicin and Cytarabine Treatment of AML Younger Patients
Acronym: FAMYLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAMYLY
Record Dates: First submitted 2013-11-15; First posted 2013-12-03 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML; high-risk cytogenetics; younger patients; Induction treatment; OMEGAVEN
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fish oil triglycerides; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OMEGAVEN - Daunorubicin - Cytarabine (Experimental): If WBC ≥ 30 G/L, chemotherapy the induction cycle :
  * Daunorubicin 60 mg/m²/day IV on D1, D2, and D3
  * Cytarabine 200 mg/m²/day D1 to D7
  * OMEGAVEN® 2 ml/kg D1 to D9,
  If WBC ≤ 30 G/L, OMEGAVEN during 48 hours
  Induction cycle :
  OMEGAVEN® 2 ml/kg D-2 to D7 Daunorubicin 60 mg/m²/day IV on D1, D2, and D3
  - Cytarabine 200 mg/m²/day IV D1 to D7
  bone marrow aspirate at D15: If BM blasts are > 5% or if second induction course :
  * Daunorubicin 35 mg/m²/day IV D17 and D18
  * OMEGAVEN® 2 ml/kg
  * Cytarabine 1000 mg/m²/12h IV on D17, D18, and D19
  For all patients: G-CSF 5 µg/kg/day subcutaneously from D21 to hematopoietic recovery (PMN > 1 G/L or > 0.5 G/L during 3 days).
  Consolidation will be administered at investigator's discretion
  Interventions: Drug: OMEGAVEN; Drug: Daunorubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: OMEGAVEN — AML Study treatment induction phase
Drug: Daunorubicin — AML Study treatment induction phase
  Other Names: Cerubidine
Drug: Cytarabine — AML Study treatment induction phase
  Other Names: Aracytine

SUMMARY:
Pilot study of the efficacy and tolerance of the adjunction of a Fish oil emulsion to daunorubicin and cytarabine chemotherapy for the treatment of Acute MYeloblastic Leukemia of Younger patients (under 61 years) with high-risk cytogenetics.

DETAILED DESCRIPTION:
Adjunction of a Fish oil emulsion OMEGAVEN to daunorubicin and cytarabine chemotherapy for the treatment of Acute MYeloblastic Leukemia of Younger patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 60 years old (less than 61 years old)
* With newly diagnosed with AML according to WHO classification:
* With 20% or more blasts in the bone marrow
* Patients with history of tumors other than myeloproliferative disorders or myelodysplastic syndromes, having received chemotherapy and/or radiotherapy without previous history of myelodysplastic syndromes are eligible for the present study
* High-risk cytogenetics defined as one the following abnormalities : 5/5q-, 7/7q-, t(6,9), 11q23 abnormality excluding t(9;11), 3q abnormality,complex karyotype (>3 abnormalites)
* Left ventricular ejection fraction (LVEF) > 50% on echocardiography or multigated acquisition (MUGA) scan or similar radionuclide angiographic scan.
* Adequate liver function (all of the following) except if secondary to the leukemia:

Total bilirubin below 1.5 x upper limit of normal (ULN), AST and ALT below 2.5 x ULN , gamma-GT below 2.5 x ULN,

* Adequate kidney function (all of the following): Serum creatinine below 1.5 x ULN, Creatinine clearance above 50 mL/min (Cockroft and Gault formula)
* ECOG performance status < or = 2.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* The patient must give written (personally signed and dated) informed consent before completing any study-related procedure which means assessment or evaluation that would not form part of the normal medical care of the patient.
* Affiliated to the French Social Security (Health Insurance).

Exclusion Criteria:

* Previous allogeneic stem cell transplantation.
* Pre-existing aplastic anemia
* Presence of favourable cytogenetics with t(8;21), t(15;17), or inv(16)
* Previous history of MDS or myeloproliferative neoplasm
* Uncontrolled active infection.
* History of arrythmia.
* Cardiac toxicity induced by another anthracycline administration
* Maximum cumulative dose reached for any anthracyclin
* Allergy to cytarabine, daunorubicin, fish or egg proteins10. Significant neurologic (grade > 2) or psychiatric disorder, dementia or seizures.
* Clinical symptoms suggesting active central nervous system leukemia.
* Degenerative or toxic encephalopathy
* Severe complications of leukemia such as:Uncontrolled bleeding, Pneumonia with hypoxia or shock
* Prior total body irradiation > 10 Gy.
* Known active HIV, Hepatitis B or C infection
* Pregnancy or breastfeeding
* Concomitant anti-amarile vaccination (yellow fever)
* Concurrent treatment with any other anti-cancer therapy except Hydroxyurea

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
response to study treatment | 1 month
  Number of patients incomplete response rate after the adjunction of a Fish oil emulsion to daunorubicin and cytarabine chemotherapy for the induction of untreated AML

SECONDARY OUTCOMES:
Tolerance | 4 months
  Number of patients with side effects during and after the admistration of a Fish oil emulsion with daunorubicin and cytarabine chemotherapy for the induction of untreated AML
Efficacy on peripheral blasts decrease | 1 month
  Daily quantification of peripheral blasts by flow cytometry during the adjunction of a Fish oil emulsion to daunorubicin and cytarabine chemotherapy
pharmacokinetics | 1 month
  Measure of plasma concentration of daunorubicin and cytarabine administered together with a fish oil emulsion

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel GYAN, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Emmanuel GYAN, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gyan E, Pigneux A, Hunault M, Peterlin P, Carre M, Bay JO, Bonmati C, Gallego-Hernanz MP, Lioure B, Bertrand P, Vallet N, Ternant D, Darrouzain F, Picou F, Bene MC, Recher C, Herault O. Adjunction of a fish oil emulsion to cytarabine and daunorubicin induction chemotherapy in high-risk AML. Sci Rep. 2022 Jun 13;12(1):9748. doi: 10.1038/s41598-022-13626-y. PMID 35697729
- [Derived] Picou F, Debeissat C, Bourgeais J, Gallay N, Ferrie E, Foucault A, Ravalet N, Maciejewski A, Vallet N, Ducrocq E, Haddaoui L, Domenech J, Herault O, Gyan E. n-3 Polyunsaturated fatty acids induce acute myeloid leukemia cell death associated with mitochondrial glycolytic switch and Nrf2 pathway activation. Pharmacol Res. 2018 Oct;136:45-55. doi: 10.1016/j.phrs.2018.08.015. Epub 2018 Aug 22. PMID 30142422
- [Derived] Gyan E, Raynard B, Durand JP, Lacau Saint Guily J, Gouy S, Movschin ML, Khemissa F, Flori N, Oziel-Taieb S, Bannier Braticevic C, Zeanandin G, Hebert C, Savinelli F, Goldwasser F, Hebuterne X; NutriCancer2012 Investigator Group. Malnutrition in Patients With Cancer: Comparison of Perceptions by Patients, Relatives, and Physicians-Results of the NutriCancer2012 Study. JPEN J Parenter Enteral Nutr. 2018 Jan;42(1):255-260. doi: 10.1177/0148607116688881. Epub 2017 Dec 11. PMID 29505137
- See also: FILO site — http://www.filo-leucemie.org